CLINICAL TRIAL: NCT06430528
Title: A Block-and-Replace Therapy With Osilodrostat and Concomitant Glucocorticoid Replacement
Status: Recruiting | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: RECORDATI GROUP (Industry)
Responsible Party: Principal Investigator, Richard J. Auchus, MD PhD, Professor of Translational Medicine, Professor of Internal Medicine and Professor of Pharmacology, University of Michigan
Other Study IDs: HUM00246263
Record Dates: First submitted 2024-04-24; First posted 2024-05-28 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Endogenous Cushing Syndrome; Adrenal Insufficiency; Hypercortisolism
Keywords: Osilodrostat; Glucocorticoid; Methylprednisolone; Medrol
MeSH Terms: conditions — Adrenal Insufficiency; Cushing Syndrome | interventions — Osilodrostat

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples for steroid measurements.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational cohort: Participants with Cushing syndrome consented to participate in block-and-replace osilodrostat therapy.
  Interventions: Drug: Osilodrostat

INTERVENTIONS:
Drug: Osilodrostat — Add methylprednisolone to osilodrostat therapy after first dose and continue during osilodrostat titration.
  Other Names: Isturisa

SUMMARY:
The major goal of this study is to determine the incidence of adrenal insufficiency in patients with endogenous Cushing syndrome receiving osilodrostat treatment combined with a replacement of glucocorticoid (block-and-replace approach).

The investigators are also evaluating new biomarker steroids to reflect adequate osilodrostat dosing, the durability and safety, and clinical improvement during treatment.

DETAILED DESCRIPTION:
Phase 1 (Titration):

Participants will provide written informed consent and receive the first dose of osilodrostat (1-2 mg) in the evening. The following morning, participants will add treatment with at least a physiologic replacement dose of methylprednisolone (4-6 mg/d based on body size in not more than 2 divided doses) and concurrently continue 1-2 mg BID of osilodrostat. Frequent communication is maintained with each participant, at least twice weekly for the first 3 months and weekly thereafter until target osilodrostat dose is reached. Study personnel will ask targeted questions related to the primary endpoint with parameters to notify the study physicians for early signs of adrenal insufficiency. Participants are instructed to double their methylprednisolone dose for intercurrent illness and for symptoms of cortisol deficiency or withdrawal that do not resolve with pausing osilodrostat dosing. Every 4-12 weeks, an AM cortisol, as well as a research sample for steroid profiling (including 11OHA4), is obtained prior to the first doses of methylprednisolone and osilodrostat. The osilodrostat dose is up-titrated as necessary to achieve an AM cortisol goal of <5 µg/dL. Once the AM cortisol is at goal, a late-night saliva cortisol (LNSC) and 24 h urine free cortisol (UFC) is obtained per standard of care. Osilodrostat titration is continued if necessary until the UFC is also at goal of <10 µg/24h. Once the AM cortisol and UFC are at goals (<5 µg/dL and <10 µg/24h, respectively), the primary endpoint measures are completed, and the participant enters Phase 2.

Phase 2 (Maintenance):

Once the participant reaches what the investigator considers the maintenance doses of osilodrostat and methylprednisolone, participants are followed for a total of 48 weeks from the first osilodrostat dose before being considered at the end of study. The AM serum cortisol, UFC, and LNSC are repeated at the end of the 48-week period and as clinically indicated throughout Phase 2, generally every 3-6 months.

ELIGIBILITY:
Inclusion Criteria:

* Endogenous Cushing syndrome, either following surgery or not candidates for surgery
* Under consideration to receive osilodrostat as part of their clinical care
* Able to provide informed consent.

Exclusion Criteria:

* Treatment with other investigational drugs within 30 days or five half-lives (whichever is longer).
* A history of hypersensitivity to osilodrostat or therapies of a similar chemical class.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving care at the University of Michigan.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2024-07-19 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Percent of participants who experience an adrenal insufficiency event during Phase 1 (titration phase) | Through phase 1, approximately 24 weeks
  based on evidence of hypotension (systolic BP <90 mmHg) and/or hypoglycemia (glucose <45 mg/dL) with antecedent symptoms (examples: anorexia, nausea, abdominal pain, orthostasis) and with a resolution of signs upon receiving rescue glucocorticoid therapy

SECONDARY OUTCOMES:
Correlation between AM cortisol and 11OHA4 measurements | Up to end of study, approximately 48 weeks
  compare biomarkers measured by mass spectrometry. This may be calculated Upon 12 participants completing phase 1 or at the end of the study, whichever comes first.
Rate of adrenal insufficient episodes per patient per year | Up to end of phase 2 (approximately 48 weeks)
  based on evidence of hypotension (systolic BP <90 mmHg) and/or hypoglycemia (glucose <45 mg/dL) with antecedent symptoms (examples: anorexia, nausea, abdominal pain, orthostasis) and with a resolution of signs upon receiving rescue glucocorticoid therapy
Frequency of cortisol withdrawal symptoms | Up to end of phase 2 (approximately 48 weeks)
  Based on patient-reported outcomes
Change in weight | Baseline, end of phase 2 (approximately 48 weeks)
  Based on clinic measurements
Change in diastolic blood pressure | Baseline, end of phase 2 (approximately 48 weeks)
  Based on clinic measurements
Change in systolic blood pressure | Baseline, end of phase 2 (approximately 48 weeks)
  Based on clinic measurements
Mean change in HgbA1c for participant with HgbA1c > 6.4% at entry. | Baseline, end of phase 2 (approximately 48 weeks)
  Based on clinic measurements
Change in number of concomitant medications | Baseline, end of phase 2 (approximately 48 weeks)
  Based on clinic notes, total number of medications used to treat Cushing syndrome comorbidities
Adrenal Insufficiency Assessment Questionnaire scores | Up to end of study, approximately 48 weeks
  Custom questionnaire for adrenal insufficiency- 4 Likert questions with scores ranging from 4-20. Higher scores indicate worse symptoms.
RAND Short Form (SF)-36 scores | Up to end of study, approximately 48 weeks
  The 36-Item Short Form Health Survey (SF-36) is standard RAND form used clinically. It is a set of generic, coherent, and easily administered quality-of-life measures. Scores for the scale range from 0-100 with higher scores indicating a better Health-related Quality of Life.
Ease of titration | Up to end of phase 1 (approximately 48 weeks)
  Investigators' judgment (1-5 scale)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Auchus, MD, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No